CLINICAL TRIAL: NCT02591550
Title: A Study on the Mechanism of Cough Hypersensitivity
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Kefang Lai (Other)
Responsible Party: Sponsor-Investigator, Kefang Lai, Professor, The First Affiliated Hospital of Guangzhou Medical University
Organization: The First Affiliated Hospital of Guangzhou Medical University (Other)
Other Study IDs: coughlongli
Record Dates: First submitted 2015-10-21; First posted 2015-10-29 (Estimated); Last update posted 2015-10-29 (Estimated); Status verified 2015-10

CONDITIONS: Cough
Keywords: chronic cough; cough reflex sensitivity; transient receptor potential vanilloid 1; transient receptor potential ankyrin 1
MeSH Terms: conditions — Cough; Chronic Cough

STUDY DESIGN:
Observational Model: Case-Control
Biospecimen Retention: Samples Without DNA — mucosa of upper trachea
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- patients with normal cough sensitivity
- patients with high cough sensitivity
- healty controls

SUMMARY:
The aim of this study is described as follows,

1. To establish a validated method to test cough reflex sensitivity conducted by transient receptor potential vanilloid 1(TRPV1).
2. To observe the variance of cough reflex sensitivity conducted by transient receptor potential ankyrin 1(TRPA1) of chronic patients and the relationship between cough reflex sensitivity conducted by TRPA1 and conducted by TRPV1.
3. To study the distribution of TRPA1 and TRPV1 channels and their relationship to cough reflex sensitivity.

DETAILED DESCRIPTION:
This study is divided into two major part, Firstly,to observe the variance of cough reflex sensitivity of chronic cough patients and the relationship between it and airway inflammation.

1. Recruit chronic cough patients and healthy volunteers as subjects.
2. Help subjects to complete detailed history,physical examination,Hull airway reflux questionnaire,chest x-rays,induced sputum,blood routine test,pulmonary ventilation function test and histamine provocation test before they enter this study.
3. Complete allyl isothiocynate(AITC) cough provocation test the day subjects enter the study,then complete capsaicin（CAP）cough provocation test after 3 days.
4. To detect the substance P(SP),calcitonin gene-related peptide(CGRP),prostaglandin E2(PGE2),et al level in sputum supernatants.

Secondly,to observe the distribution of TRPA1,TRPV1 channels and the relationship between it and cough reflex sensitivity.

1）Recruit chronic cough patients and healthy volunteers and complete related examinations as mentioned before.

2)Collect mucosa specimens from upper trachea via endobronchial biopsy,and airway epithelial cells from 2nd or 3rd order bronchi via brushing.

3)Evaluate the expression level of TRPA1,TRPV1 of mucosa specimens of subjects by immunofluorescent assay and Image analysis software.

4)Cultivate airway epithelial cells from subjects and evaluate the expression of TRPV1,TRPA1 and functional changes of it.

ELIGIBILITY:
Inclusion Criteria:

chronic cough group:

1. cough lasting ≥ 8 weeks,characterized by irritating dry cough.
2. sensitive to fumes，dust,the odorous and cold air.
3. with normal chest x-rays. 4.17-70 years old.

5.without smoking history. healty controls group: 1.17-70 years old. 2.without smoking hitory or stop smoking for more than 2 years. 3.without chronic cough. 4.without chronic respiratory diseases. 5.without chronic heart, liver, kidney,and autoimmune disease. 6.with normal chest x-rays. 7.with normal pulmonary ventilation function,and histamine challenge test showed negative result.

Exclusion Criteria:

chronic cough group and healty controls group:

1. with respiratory tract infection within 8 weeks.
2. with chronic respiratory diseases or severe heart, liver, kidney,and autoimmune disease.
3. using Angiotensin-Converting Enzyme Inhibitors(ACEI),bronchodilators,glucocorticosteroid,antihistaminics within one week.
4. women during pregnancy or lactation.
5. patients with malignant tumours.

Ages: 17 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Chronic cough group:nonsmokers with chronic cough lasting ≥ 8 weeks characterized by irritating dry cough or small amount of sputum, sensitive to fumes，dust, cold air ,and normal chest x-ray were enrolled.
  Healthy control:healthy volunteers presented our hospital for healthy examination were enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2015-03; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
TRPA1,TRPV1 channels expression level of chronic cough patients and its relationship with cough reflex sensitivity | 7 days post-bronchoscopy
  Complete AITC cough provocation test the day subjects enter the study,then complete CAP cough provocation test after 3 days,record the threshold of cap and aitc concentration(mmol/L) when it cause subjects cough equal to or more than 5 times.Measure the expression level of TRPA1 and TRPV1 of biopsy sample from chronic cough patients and healthy controls by immunofluoresent assay 7 days post bronchoscopy.Analyze the statistic by spss18.0.

SECONDARY OUTCOMES:
The relationship between CAP cough reflex sensitivity test conducted by TRPV1 and AITC cough reflex sensitivity test conducted by TRPA1 | 7 days post-bronchoscopy
  Complete AITC cough provocation test the day subjects enter the study,then complete CAP cough provocation test after 3 days,record the threshold of cap and aitc concentration(mmol/L) when it cause subjects cough equal to or more than 5 times.Analyze the statistic by spss18.0.

CONTACTS AND LOCATIONS:
Locations (1):
- Guangzhou Institute of Respiratory Disease, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Lai K, Long L, Yi F, Tang J, Chen Z, Chen F, Zhou J, Peng W, Zhang L, Li H, Zhan W, Chen R, Luo W, Chen Q, Chung KF, Zhong N. Age and Sex Distribution of Chinese Chronic Cough Patients and Their Relationship With Capsaicin Cough Sensitivity. Allergy Asthma Immunol Res. 2019 Nov;11(6):871-884. doi: 10.4168/aair.2019.11.6.871. PMID 31552721
- [Derived] Long L, Yao H, Tian J, Luo W, Yu X, Yi F, Chen Q, Xie J, Zhong N, Chung KF, Lai K. Heterogeneity of cough hypersensitivity mediated by TRPV1 and TRPA1 in patients with chronic refractory cough. Respir Res. 2019 Jun 6;20(1):112. doi: 10.1186/s12931-019-1077-z. PMID 31170994